CLINICAL TRIAL: NCT02225756
Title: Brief Administration of Cyclosporine A to Induce the Stabilisation of the Diameter of Small Diameter Abdominal Aortic Aneurysms.
Brief Title: Cyclosporine A in Patients With Small Diameter Abdominal Aortic Aneurysms
Acronym: ACA4
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P110119
Record Dates: First submitted 2014-08-06; First posted 2014-08-26 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Abdominal Aortic Aneurysm,; Small Abdominal Aortic Aneurysm
Keywords: Drug therapy; Prevention and control; Healing; Tissue regeneration; Therapy
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cyclosporine A dose 1 (Experimental)
  Interventions: Drug: Cyclosporine A
- Cyclosporine A dose 2 (Experimental)
  Interventions: Drug: Cyclosporine A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine A — Oral administration for a short time of cyclosporine A dose 1
  Arms: Cyclosporine A dose 1
Drug: Cyclosporine A — Oral administration for a short time of cyclosporine A dose 2
  Arms: Cyclosporine A dose 2
Drug: Placebo — Oral administration for a short time of placebo
  Arms: Placebo

SUMMARY:
Aneurysms of the aorta are dilatations of the main artery in the body that distributes blood to organs. Aneurysms expose patients to aortic rupture. The risk of aortic rupture is high for large aneurysms, and low for small aneurysms. Currently, if the diameter of a small aneurysm grows up to a level at risk for rupture, surgery is indicated to prevent rupture. A drug that would stop growth of small aneurysms would obviate aortic surgery, the current treatment to prevent aortic rupture in patients. The ACA4 study aims at testing the possibility to stop growth of small aortic aneurysms in the abdomen with a drug, cyclosporine A. Patients with small aneurysms will receive cyclosporine A orally, or a placebo (fake liquid), every day during a short period of time. Efficacy of the drug will be evaluated by measuring the diameter of the aneurysm during 2 years after treatment cessation. Drug safety analysis will evaluate the impact of the drug on renal function, blood pressure, and other parameters. In case of adverse event during the drug administration phase, dose of the drug or of the placebo will be decreased or administration stopped.

DETAILED DESCRIPTION:
Abdominal aortic aneurysms (AAAs) expose patients to death caused by aortic rupture. Although screening of AAAs has been shown to decrease AAA-related mortality, translation into medical practice of screening is limited because there is no specific treatment to limit growth of AAAs below diameter thresholds for open surgery or stent graft. We have developed different approaches aimed at inducing healing and thereby stabilizing formed AAAs in animal models. We have identified TGF-beat1 as an inducer of experimental AAA healing. Cyclosporine A is an inducer of tumor growth factor - beta1 (TGF-beta1) in experimental AAAs and in human atherosclerotic AAAs in vitro, causing overgrowth of inflamed tissues. Since AAAs are caused by aortic wall atrophy, we have hypothesised and confirmed in animals, that cyclosporine AAA, when administrated during a short period of time, durably stabilizes small AAA diameter in animals, while inducing aortic wall reconstruction and healing.

The clinical trial ACA4 is a multicentric randomized, placebo controlled, double blind trial that will enrol 360 patients with small AAAs in France. Two doses of cyclosporine A will be tested against a placebo (three arms). Drug administration will be short, and AAA diameter evaluation will be performed for 2 years, by CT-scanner (main outcome) with no contrast, and duplex-scanner.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with asymptomatic AAA ≥ 30 mm, ≤ 49 mm
* Female patients with asymptomatic AAA ≥ 25 mm, ≤ 44 mm

Exclusion Criteria:

* Common iliac aneurysm > 25 mm
* Saccular aneurysm of the aorta
* Inflammatory aneurysm
* No signature of informed consent
* Renal dysfunction
* Diabetes

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
AAA diameter evolution on CT-scanner 12 months after treatment interruption | 1 years

SECONDARY OUTCOMES:
AAA diameter evolution on duplex-scanner 12 months after treatment interruption | 1 years
Renal function (creatinine clearance) | at inclusion visit, V4 and V8
All cause cardiovascular mortality and morbidity | at V1 and V8

CONTACTS AND LOCATIONS:
Overall Officials: Eric Allaire, MD. PhD., Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France